CLINICAL TRIAL: NCT01683318
Title: Thermal Pulsation System for the Treatment of Meibomian Gland Dysfunction
Brief Title: Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R913/22/2012
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2012-09

CONDITIONS: Meibomian Gland Dysfunction (MGD)
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients will undergo Thermal Pulsation treatment of Meibomian Gland Dysfunction using the TearScience System (Lipiflow).
  Interventions: Procedure: Thermal Pulsation therapy

INTERVENTIONS:
Procedure: Thermal Pulsation therapy

SUMMARY:
The current study aims to test the efficacy of treatment for a device that utilises a thermal pulsation system, which applies heat from the inner surface of the eyelids (Lipiflow) in patients suffering from meibomian gland dysfunction.

Patients will be asked to undergo a one-time treatment with Lipiflow and the investigators will monitor them for changes in tear film and lipid composition, as well as changes in the anatomy of meibomian glands for over a study period of 12 weeks. Additionally, dry eye symptoms will be documented in form of questionnaires.

The investigators hypothesize that the treatment will be effective in improving clinical signs and will relieve dry eye symptoms for the patient. If this method of managing Meibomian Gland Dysfunction (MGD) is found to be efficacious and safe, it will be made available to patients in Singapore.

ELIGIBILITY:
Inclusion Criteria:

1. Eyelids must present with blocked meibomian gland openings (plugs), at least 1 visible MG plug in the 4 eyelids, or discernable change in consistency of meibum (increased in viscosity or opacity) when MG expressed in upper or lower eyelids.
2. At least one out of 8 questions on dry eye symptoms is answered with often or all the time.
3. Eyes should not show any other ocular surface pathology which required more treatment than eye lubricant and conventional eyelid hygiene.

Exclusion Criteria:

1. Known history of thyroid disorders (diagnosed by physician).
2. No ocular surgery within the previous 6 months and LASIK within the previous 1 year.
3. Any intake of central nervous system and hormonal drugs within last 30 days and inability to withhold such drugs for at least 6 weeks.
4. Active ocular infection or pterygium.
5. Anticipated necessity to wear contact lens in the duration of the study.
6. Living in the same household as another participant of the study.
7. Any other specified reason as determined by clinical investigator, for example, the need to use any treatment or eyedrops not permitted by the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
ocular discomfort | 3 months

SECONDARY OUTCOMES:
Tear Break Up Time (TBUT) | 3 months
Number of blocked meibomian glands | 3 months
Corneal fluorescein staining score | 3 months
To measure the production of tears | 3 months
  Schirmer's test uses paper strips inserted into the lower eyelid (conjunctival sac)for 5 minutes to measure the production of tears. Both eyes are tested at the same time. The paper is then removed and the amount of moisture is measured.
Tear evaporimetry | 3 months
Lipid layer thickness | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Yeo S, Tan JH, Acharya UR, Sudarshan VK, Tong L. Longitudinal Changes in Tear Evaporation Rates After Eyelid Warming Therapies in Meibomian Gland Dysfunction. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(4):1974-81. doi: 10.1167/iovs.16-19088. PMID 27096755